CLINICAL TRIAL: NCT02555488
Title: Comparing the Antibacterial Effect of 810 nm Diode Laser and Photodynamic Therapy in Reducing the Microbial Flora of the Canal While Root Retreatment in Patients With Periradicular Lesions
Brief Title: Comparing the Antibacterial Effect of 810 nm Diode Laser and Photodynamic Therapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University (Other)
Responsible Party: Principal Investigator, saranaz azari-marhabi, dr, Shahid Beheshti University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: shahid beheshti university
Record Dates: First submitted 2015-09-15; First posted 2015-09-21 (Estimated); Last update posted 2015-09-21 (Estimated); Status verified 2015-09

CONDITIONS: Periradicular Disease
MeSH Terms: conditions — Periapical Diseases | interventions — Lasers, Semiconductor; Methylene Blue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Experimental): in the second group diode laser (810 nm, 1.2 W, 30 s) was irradiated. Then second samples were taken from all canals.
  Interventions: Device: diode laser
- 1 (Experimental): In the first group Photodynamic therapy (PDT) with Methylene blue and diode laser (810 nm, 0.2 W, 40 second) was done
  Interventions: Device: diode laser; Drug: Methylene blue

INTERVENTIONS:
Device: diode laser — MB and diode
  Arms: 1
Device: diode laser — diode laser
  Arms: 2
Drug: Methylene blue — Methylene blue and diode laser was used
  Arms: 1

SUMMARY:
The aim of this study was to compare the Antibacterial Efficacy of Diode Laser 810nm and Photodynamic therapy in reducing bacterial microflora in endodontic retreatment of teeth with periradicular lesion.

DETAILED DESCRIPTION:
Conventional techniques of root canal treatments such as mechanical instrumentation and chemical debridement with antimicrobial irrigants, such as Sodium hypochlorite (NaOCl) and chlorhexidine and use of calcium hydroxide do not always suffice to predictably render root canals free of bacteria Using the high-power diode laser is a new approach of disinfection allowing access to the previously unavailable areas, such as the tubular network. This study, therefore, compares two types of diode lasers (low-power and high power) in terms of anti-bacterial effect as well as the conventional endodontic retreatment to determine the ideal method of root canal disinfection.

ELIGIBILITY:
Inclusion Criteria:

- endodontic retreatment of teeth with periradicular lesion.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-10 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
bacterial colony forming unit(CFU/ML) | 12 months
  after doing protocol in each groups CFU /ml for different bacteria will be counted

CONTACTS AND LOCATIONS:
Overall Officials: saranaz azari-marhabi, DMD, Principal Investigator — Shahid Beheshti University of Medical Sciences
Locations (1):
- Shahid Beheshti University, Tehran, Iran